CLINICAL TRIAL: NCT01458522
Title: Utility of Intravenous Lacosamide Compared With Fosphenytoin in the Treatment of Patients With Frequent Nonconvulsive Seizures
Brief Title: Intravenous Lacosamide Compared With Fosphenytoin in the Treatment of Patients With Frequent Nonconvulsive Seizures
Acronym: TRENdS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aatif Husain (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor-Investigator, Aatif Husain, MD, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00033295; Pro00037794 (Other: Duke Site Protocol Number); DCRI-CEMC101.01
Record Dates: First submitted 2011-10-20; First posted 2011-10-25 (Estimated); Results first posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Nonconvulsive Seizures
Keywords: Nonconvulsive Seizures
MeSH Terms: interventions — fosphenytoin; Lacosamide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fPHT 20mg (Active Comparator): fPHT treatment arm, a bolus of 20 mg PE/kg will be administered at a rate of no greater than 75 mg PE/minute. If a further bolus is required, 5 mg PE/kg will be administered. The daily maintenance dose for fPHT will be 5 mg PE/kg divided into 2 doses.
  Interventions: Drug: fPHT; Drug: LCM
- LCM 400mg (Experimental): LCM treatment arm, a bolus of 400 mg will be administered over 30 minutes. If a further bolus is required, 200 mg will be administered. Regardless of whether the subject received a rebolus, he or she will begin receiving a maintenance dose 12 hours after the initial dose. The daily maintenance dose will be the same as the total bolus (400 mg or 600 mg) divided into 2 doses.
  Interventions: Drug: fPHT; Drug: LCM

INTERVENTIONS:
Drug: fPHT — If after initial treatment with fPHT any of the following occurs, the subject will have reached the end of the first treatment arm and will "cross over" and begin receiving the other drug, ie, the one not originally administered: the subject subsequently has another seizure within 24 hours following the 2-hour post-rebolus observation-only period; the subject does not receive a rebolus but has a seizure within 24 hours following the 2 hour post-bolus observation-only period; the subject experiences an AE that precludes further use of the first study drug.
  If crossover occurs, the subject will "start over" with the second drug, going through the same observation-only period, rebolusing (if necessary), and study assessments with the second drug, beginning with the Baseline assessments.
  Other Names: Cerebyx, Fosphenytoin
Drug: LCM — If after initial treatment with LCM any of the following occurs, the subject will have reached the end of the first treatment arm and will "cross over" and begin receiving the other drug, ie, the one not originally administered: the subject subsequently has another seizure within 24 hours following the 2-hour post-rebolus observation-only period; the subject does not receive a rebolus but has a seizure within 24 hours following the 2 hour post-bolus observation-only period; the subject experiences an AE that precludes further use of the first study drug.
  If crossover occurs, the subject will "start over" with the second drug, going through the same observation-only period, rebolusing (if necessary), and study assessments with the second drug, beginning with the Baseline assessments.
  Other Names: Vimpat, Lacosamide

SUMMARY:
This a phase 2 study comparing the efficacy of intravenous (IV) lacosamide (LCM) with IV fosphenytoin (fPHT) in controlling frequent nonconvulsive seizures (NCSs), the Adverse Events profile of LCM compared with fPHT when used to treat frequent NCSs, and length of stay in an intensive care unit for subjects treated with LCM versus subjects treated with fPHT. The trial will include a preacute-treatment period, an acute-treatment period, a postacute-treatment period, and a long-term follow-up period.

DETAILED DESCRIPTION:
Exploratory, prospective, multicenter, open-label, randomized study, in which the physicians who are interpreting cEEGs for treatment purposes and the central reviewers who are providing final cEEG interpretation for study purposes are all blinded to treatment.

Initial LCM/maintenance doses: Subjects will receive a 400-mg IV initial bolus over 30 minutes, followed by a 2-hour post-dose observation-only period. If a breakthrough seizure occurs in the 6 hours following the 2-hour post-dose observation-only period, the subject will receive a 200-mg rebolus over 30 minutes. Regardless of whether a rebolus was administered, a maintenance dose of LCM will be started 12 hours after the initial bolus, and it will continue every 12 hours throughout the acute-treatment period. The daily maintenance dose will be equivalent to the total IV bolus per day (400 mg if no rebolus was administered or 600 mg if a rebolus was administered), divided into 2 doses. After completion of the acute-treatment period, daily maintenance with an AED will be at the discretion of the treating physician.

Initial fPHT/maintenance doses: Subjects will receive a 20-mg PE/kg IV initial bolus at a rate no greater than 75 mg PE/minute, followed by a 2-hour post-dose observation-only period. If a breakthrough seizure occurs in the 6 hours following the 2-hour post-dose observation-only period, the subject will receive a 5-mg PE/kg IV rebolus at a rate no greater than 75 mg PE/minute. Regardless of whether a rebolus was administered, a maintenance dose of fPHT will be started 12 hours after the initial bolus, and it will continue every 12 hours throughout the acute-treatment period. The daily maintenance dose will be 5 mg PE/kg, divided into 2 doses. After completion of the acute-treatment period, daily maintenance with an AED will be at the discretion of the treating physician.

Crossover/maintenance doses: If a subject does not receive a rebolus but has a seizure within 24 hours following the 2-hour post-initial-dose observation-only period, he or she will "cross over" and begin receiving the other drug, ie, the one not originally administered. If a subject does receive a rebolus and has another seizure within 24 hours following the 2-hour post-rebolus observation-only period, he or she will also cross over to the other drug. If crossover occurs, the subject will "start over" with the second drug, going through the same observation-only period and rebolusing, if necessary. If a subject crosses over and starts receiving the second drug, in addition to receiving every-12-hours maintenance doses of the drug originally administered, the subject will also receive maintenance doses of the second drug every 12 hours, beginning 12 hours after the first dose of the second drug.

ELIGIBILITY:
Inclusion Criteria:

1. Have the capacity to understand and sign an institutional review board (IRB)-approved informed consent form (ICF) or have a legally authorized representative (LAR) available to sign on behalf of the subject.
2. Are undergoing cEEG monitoring in the neurologic intensive care unit (NICU) or other closely monitored environment.
3. Are experiencing NCSs according to the following criteria:

   * At least 1 ESz lasting at least 10 seconds, with or without clinical correlates, occurring within the last 6 hours of cEEG monitoring.
   * If a new AED has been started, ESzs must have occurred per the preceding bullet point at least 2 hours after starting that AED.
   * If individual ESzs are not well defined, ESz time is at least 10 seconds and less than 30 minutes per hour of cEEG recording.
4. Are being considered for treatment with an IV AED.
5. Are at least 18 years old.

Exclusion Criteria:

1. Treatment with PHT, fPHT, or LCM in the last 7 days.
2. Contraindication for the use of fPHT or LCM.
3. Ongoing generalized convulsive status epilepticus (SE) (more than 2 generalized tonic-clonic seizures within 30 minutes without recovery to baseline or 1 seizure lasting longer than 10 minutes).
4. Episodes of SE, defined as at least 30 minutes of ESz activity in 1 hour, in the last 6 hours.
5. Encephalopathic event secondary to acute anoxic/hypoxic event.
6. Undergoing therapeutic hypothermia protocol.
7. Continuous EEG monitoring showing only periodic discharges or rhythmic delta activity without clear ESzs (for definitions of periodic discharges, rhythmic delta activity, and ESzs, see the Manual of Operations).
8. Electroencephalographic seizures consistent with typical absence seizures.
9. Evaluation for spell characterization or surgical treatment for epilepsy.
10. Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aatif Husain, MD, Principal Investigator — Duke Clinical Research Institute
Locations (11):
- United States (11):
  - Huntington Memorial Hospital, Pasadena, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Emory University School of Medicine, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Woman's Hospital, Boston, Massachusetts
  - Mission Hospital, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center Dallas, Dallas, Texas

REFERENCES:
- [Derived] Belcastro V, Vidale S, Pierguidi L, Sironi L, Tancredi L, Striano P, Taborelli A, Arnaboldi M. Intravenous lacosamide as treatment option in post-stroke non convulsive status epilepticus in the elderly: a proof-of-concept, observational study. Seizure. 2013 Dec;22(10):905-7. doi: 10.1016/j.seizure.2013.07.011. Epub 2013 Aug 13. PMID 23953988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 173 participants consented. 74 participants were randomized.
Pre-assignment Details: 37 participants randomized to LCM, however 2 participants did not receive drug. 37 participants were randomized to fPHT and everyone received drug.
Groups:
- LCM First, Then fPHT: LCM bolus of 400 mg administered over 30 minutes. If further bolus is required, 200 mg is administered. Regardless of whether the subject received a rebolus, they will begin receiving a maintenance dose 12 hrs after initial dose. Daily maintenance dose will be the same as the total bolus (400 mg or 600 mg) divided into 2 doses.
  If after initial treatment and any of the following occurs, subject will have reached end of 1st treatment arm and will crossover and receive the other drug. If any of the following did not occur the subject will be considered completed.
  Subject has another seizure within 24 hrs following the 2-hr post-rebolus observation-only period.
  Subject dose not receive a rebolus but has a seizure within 24 hrs following 2-hr post bolus observation-only period.
  Subject experiences an AE that precludes further use of the 1st study drug. If crossover occurs, the subject will start over with the second drug, going through the same observation-only period.
- fPHT First, Then LCM: fPHT treatment arm, a bolus of 20 mg PE/kg will be administered at a rate of no greater than 75 mg PE/minute. If a further bolus is required, 5 mg PE/kg will be administered. The daily maintenance dose for fPHT will be 5 mg PE/kg divided into 2 doses.
  If after initial treatment and any of the following occurs, the subject will have reached the end of the first treatment arm and will "cross over" and begin receiving the other drug. If any of the following did NOT occur the subject will be considered completed.
  Subject has another seizure within 24 hours following the 2-hour post-rebolus observation-only period.
  Subject dose not receive a rebolus but has a seizure within 24 hours following 2-hour post bolus observation-only period.
  Subject experiences an AE that precludes further use of the first study drug.
  If crossover occurs, the subject will "start over" with the second drug, going through the same observation-only period, rebolusing (if necessary).
Period: Overall Study
Arm/Group | LCM First, Then fPHT | fPHT First, Then LCM
Started | 37 | 37
Received First Drug | 35 | 35
Crossover to Second Drug | 15 | 10
Completed (Completed all assigned intervention & observation. Not all subjects were assigned to crossover.) | 34 | 26
Not Completed | 3 | 11
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 1 | 9

BASELINE CHARACTERISTICS:
Groups:
- LCM First, Then fPHT: LCM treatment arm, a bolus of 400 mg will be administered over 30 minutes. If a further bolus is required, 200 mg will be administered. Regardless of whether the subject received a rebolus, he or she will begin receiving a maintenance dose 12 hours after the initial dose. The daily maintenance dose will be the same as the total bolus (400 mg or 600 mg) divided into 2 doses.
  If after initial treatment and any of the following occurs, subject will have reached the end of the first treatment arm and will "cross over" and begin receiving the other drug.
  Subject has another seizure within 24 hours following the 2-hour post-rebolus observation-only period.
  Subject dose not receive a rebolus but has a seizure within 24 hours following 2-hour post bolus observation-only period.
  Subject experiences an AE that precludes further use of the first study drug.
  If crossover occurs, the subject will "start over" with the second drug, going through the same observation-only period.
- fPHT First, Then LCM: fPHT treatment arm, a bolus of 20 mg PE/kg will be administered at a rate of no greater than 75 mg PE/minute. If a further bolus is required, 5 mg PE/kg will be administered. The daily maintenance dose for fPHT will be 5 mg PE/kg divided into 2 doses.
  If after initial treatment and any of the following occurs, the subject will have reached the end of the first treatment arm and will "cross over" and begin receiving the other drug.
  Subject has another seizure within 24 hours following the 2-hour post-rebolus observation-only period.
  Subject dose not receive a rebolus but has a seizure within 24 hours following 2-hour post bolus observation-only period.
  Subject experiences an AE that precludes further use of the first study drug.
  If crossover occurs, the subject will "start over" with the second drug, going through the same observation-only period, rebolusing (if necessary).
- Total: Total of all reporting groups
Arm/Group | LCM First, Then fPHT | fPHT First, Then LCM | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (12.1) | 63.4 (20.4) | 63.6 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 20 | 16 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 32 | 58
  Black or African American | 9 | 3 | 12
  Asian | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 37 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Experience no Nonconvulsive Seizures (NCS) for 24 Hours Following Treatment With LCM vs. fPHT, as Measured by Continuous Electroencephalography (cEEG) Monitoring.
Description: Percentage of subjects who experience no nonconvulsive seizures (NCS) for 24 hours (after the 2-hour observation-only period) following treatment with LCM vs. fPHT, as measured by continuous electroencephalography (cEEG) monitoring with blinded review.
Time Frame: 24 hours
Population: Data are reported for the percentage of participants without a nonconvulsive seizure event in the period prior to crossover.
Measure: Count of Participants; unit: Participants
Groups:
- fPHT 20mg PE/kg: fPHT treatment arm, a bolus of 20 mg PE/kg will be administered at a rate of no greater than 75 mg PE/minute. If a further bolus is required, 5 mg PE/kg will be administered. The daily maintenance dose for fPHT will be 5 mg PE/kg divided into 2 doses.
Arm/Group | LCM 400mg | fPHT 20mg PE/kg
Number analyzed (Participants) | 35 | 35
Participants | 19 | 22

2. Secondary Outcome: Percentage of Subjects Who Require a Rebolus of the Initial Antiepileptic Drugs (AED) to Control Nonconvulsive Seizures (NCS) in the LCM vs fPHT Arms.
Description: The percentage of subjects who require a rebolus of the initial antiepileptic drug (AED) to control nonconvulsive seizures (NCS) in the LCM vs fPHT arms.
Time Frame: 24 hours
Population: Data are reported for the percentage of participants who require a rebolus of the initial antiepileptic drugs (AED) to control nonconvulsive seizures (NCS) in the LCM vs fPHT arms in the period prior to crossover.
Measure: Count of Participants; unit: Participants
Arm/Group | LCM 400mg | fPHT 20mg PE/kg
Number analyzed (Participants) | 35 | 35
Participants | 16 | 13

3. Secondary Outcome: Number of Subjects Who Required a Second Antiepileptic Drug (AED) to Control Nonconvulsive Seizures (NCS)
Description: Number of subjects who required a second antiepileptic drug (AED) to control nonconvulsive seizures (NCS)
Time Frame: 24-26 hours
Population: Participants who crossed over to second drug
Measure: Count of Participants; unit: Participants
Arm/Group | LCM First, Then fPHT | fPHT First, Then LCM
Number analyzed (Participants) | 35 | 35
Participants | 15 | 10

4. Secondary Outcome: Seizure Burden Change From Baseline to End of Initial Treatment
Description: Absolute change in seizure time (defined as the number of minutes of electrographic seizure (ESz) activity per hour) before treatment and at the end of the first treatment arm. If less than 1 hour of recording time is available, seizure time will be extrapolated to 1 hour. The maximum amount of time that can be used to determine baseline seizure time is 6 hours.
Time Frame: Baseline, 24 hours
Population: Participants who had satisfactory EEG data (sometimes EEG leads would come off)
Measure: Mean (Standard Deviation); unit: min/hour
Arm/Group | LCM 400mg | fPHT 20mg PE/kg
Number analyzed (Participants) | 32 | 29
min/hour | -0.58 (0.950) | -0.54 (0.828)
Statistical Analysis 1: Comparison: LCM 400mg vs fPHT 20mg PE/kg; Test type: Other; p = 0.512, Poisson regression model

5. Secondary Outcome: Seizure Burden Change From Baseline to End of Crossover, Excluding Initial Treatment Arm
Description: Absolute change defined as the number of minutes of ESz activity per hour before treatment and at the end of the second treatment arm. This measure does not evaluate seizure activity in the first treatment arm. If less than 1 hour of recording time is available, seizure time will be extrapolated to 1 hour.
Time Frame: baseline, 26-68 hours
Population: participants who had satisfactory EEG data (sometimes EEG leads would come off)
Measure: Mean (Standard Deviation); unit: min/hour
Arm/Group | LCM First, Then fPHT | fPHT First, Then LCM
Number analyzed (Participants) | 11 | 9
min/hour | -0.78 (0.486) | -0.83 (0.346)

6. Secondary Outcome: Time of First Bolus to End of Seizures After Initial Treatment Arm, Time From Crossover to End of Seizures in Crossover Treatment Arm
Description: Time of first bolus to end of seizures after initial treatment arm, time from crossover to end of seizures in crossover treatment arm
Time Frame: time of first bolus to end of seizures after initial treatment arm, time from crossover to end of seizures in crossover treatment arm
Population: participants who had satisfactory EEG data (sometimes EEG leads would come off)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | LCM First, Then fPHT | fPHT First, Then LCM
Number analyzed (Participants) | 35 | 34
hours
  Initial Treatment | 8.4 (13.08) | 9.8 (11.84)
  Crossover Treatment: number analyzed (Participants) | 14 | 10
  Crossover Treatment | 8.2 (11.05) | 1.7 (3.46)

7. Secondary Outcome: Number of Predefined Adverse Events (AE) After Treatment Arm 1 Administration
Description: Number of predefined adverse events (AE) after treatment arm 1 administration. These predefined adverse events include Patients with at least one AE of interest, Cardiac disorders, investigations, suspected hypersensitivity reactions, vascular disorders, and hypotension.
Time Frame: 24 hours
Population: Patients who received treatment arm 1
Measure: Number; unit: Number of predefined AEs
Arm/Group | LCM 400mg | fPHT 20mg PE/kg
Number analyzed (Participants) | 35 | 35
Number of predefined AEs | 4 | 5

8. Secondary Outcome: Percentage of Subjects in Whom Study Drug is Withdrawn Early After Treatment With Treatment Arm 1
Description: Percentage of subjects in whom study drug is withdrawn early after treatment with treatment arm 1
Time Frame: baseline to end of treatment arm 1
Measure: Count of Participants; unit: Participants
Groups:
- LCM Treatment: LCM treatment arm, a bolus of 400 mg will be administered over 30 minutes. If a further bolus is required, 200 mg will be administered. Regardless of whether the subject received a rebolus, he or she will begin receiving a maintenance dose 12 hours after the initial dose. The daily maintenance dose will be the same as the total bolus (400 mg or 600 mg) divided into 2 doses.
  If after initial treatment and any of the following occurs, subject will have reached the end of the first treatment arm and will "cross over" and begin receiving the other drug.
  Subject has another seizure within 24 hours following the 2-hour post-rebolus observation-only period.
  Subject dose not receive a rebolus but has a seizure within 24 hours following 2-hour post bolus observation-only period.
  Subject experiences an AE that precludes further use of the first study drug.
  If crossover occurs, the subject will "start over" with the second drug, going through the same observation-only period.
- fPHT Treatment: fPHT treatment arm, a bolus of 20 mg PE/kg will be administered at a rate of no greater than 75 mg PE/minute. If a further bolus is required, 5 mg PE/kg will be administered. The daily maintenance dose for fPHT will be 5 mg PE/kg divided into 2 doses.
  If after initial treatment and any of the following occurs, the subject will have reached the end of the first treatment arm and will "cross over" and begin receiving the other drug.
  Subject has another seizure within 24 hours following the 2-hour post-rebolus observation-only period.
  Subject dose not receive a rebolus but has a seizure within 24 hours following 2-hour post bolus observation-only period.
  Subject experiences an AE that precludes further use of the first study drug.
  If crossover occurs, the subject will "start over" with the second drug, going through the same observation-only period, rebolusing (if necessary).
Arm/Group | LCM Treatment | fPHT Treatment
Number analyzed (Participants) | 35 | 35
Participants | 2 | 3

9. Secondary Outcome: Days in the Intensive Care Unit/Hospital
Description: Data was acquired in a manner consistent with determining if one treatment arm (LCM first, then fPHT versus fPHT first, then LCM) resulted in more days of hospitalization than the other over the course of the study.
Time Frame: initial bolus to end of study
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LCM First, Then fPHT | fPHT First, Then LCM
Number analyzed (Participants) | 37 | 37
days
  Days in ICU | 7.4 (8.36) | 6.5 (8.73)
  Days in hospital | 12.7 (7.63) | 12.5 (10.03)

10. Secondary Outcome: Change in Functional Status as Measured by the Functional Disability Scale at Day 7 to 9 Postrandomization and Day 30 Post-randomization in the LCM vs fPHT Arms.
Description: Change in functional status as measured by the Functional Disability Scale, using a 0-29 rating (0=w/o disability; 29=extreme vegetative state) at Day 7 to 9 postrandomization and Day 30 post-randomization in the LCM first, then fPHT versus fPHT first, then LCM arms. Data was analyzed in a manner consistent with determining if one treatment arm resulted in a greater change in functional status than the other.
Time Frame: Baseline to day 7-9, baseline to day 30
Population: participants who completed the Functional Disability Scale
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCM First, Then fPHT | fPHT First, Then LCM
Number analyzed (Participants) | 20 | 28
units on a scale
  Change from baseline to day 7-9 | -4.1 (7.64) | 0.3 (4.52)
  Change from baseline to day 30: number analyzed (Participants) | 14 | 20
  Change from baseline to day 30 | -8.5 (11.73) | -3.7 (5.01)

11. Secondary Outcome: Percentage of All Subjects Who Have Had a Seizure, Are on Antiepileptic Drug (AED) Therapy, and Are Alive/Dead at Day 30
Description: Percentage of all subjects who have had a seizure, are on antiepileptic drug (AED) therapy, and are alive and dead at day 30. Data was acquired in a manner consistent with determining if one treatment arm (LCM first, then fPHT versus fPHT first, then LCM) resulted in a greater effect on seizures, antiepileptic drug (AED) use, and survival at day 30 after the acute treatment period. The acute treatment period could range from 6 to 30 hours.
Time Frame: both acute treatment periods to 30 days
Measure: Number; unit: percentage of participants
Arm/Group | LCM First, Then fPHT | fPHT First, Then LCM
Number analyzed (Participants) | 45 | 50
percentage of participants
  any seizure within 30 days after acute tx period | 27.4 | 38.9
  AED use within 30 days after acute tx period | 82.2 | 74.0
  Died within 30 days after randomization | 15.5 | 16.0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 30 days after last dose of study drug (approximately 30-32 days)
Groups:
- All Participants Receiving LCM 400mg: Participants who receive a bolus of 400mg administered over 30 minutes. If a further bolus is required, 200mg will be administered. Regardless of whether the subject received a rebolus, he or she will begin receiving a maintenance dose 12 hours after the initial dose. The daily maintenance dose will be the same as the total bolus (400mg or 600mg) divided into 2 doses.
- All Participants Receiving fPHT 20mg PE/kg: Participants who receive a bolus of 20mg PE/kg administered at a rate no greater than 75mg PE/minute. If a further bolus is required, 5mg PE/kg will be administered. The daily maintenance dose for fPHT will be 5mg PE/kg divided into 2 doses.
Arm/Group | All Participants Receiving LCM 400mg | All Participants Receiving fPHT 20mg PE/kg
All-Cause Mortality (participants affected / at risk) | 7/45 | 8/50
Serious Adverse Events (participants affected / at risk) | 10/45 | 13/50
Other Adverse Events (participants affected / at risk) | 22/45 | 27/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants Receiving LCM 400mg (N=45) | All Participants Receiving fPHT 20mg PE/kg (N=50)
Bradycardia (Cardiac disorders) | 1 | 0
Herpes simplex encephalitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2
Cerebral hemorrhage (Nervous system disorders) | 2 | 1
Neurological decompensation (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypotension (Vascular disorders) | 2 | 2
Encephalitis viral (Infections and infestations) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants Receiving LCM 400mg (N=45) | All Participants Receiving fPHT 20mg PE/kg (N=50)
Bradycardia (Cardiac disorders) | 2 | 2
Atrial tachycardia (Cardiac disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Herpes simplex encephalitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Incorrect route of drug administration (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Heart rate abnormal (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 1
Neurological decompensation (Nervous system disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 1
rash (Skin and subcutaneous tissue disorders) | 0 | 2
hypotension (Vascular disorders) | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Encephalitis viral (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No